CLINICAL TRIAL: NCT06766305
Title: Phase Ib/II Clinical Study of QL1706 Combined With SOX Perioperative Treatment for Resectable Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: QL1706 Combined With SOX Used in Theperioperative Treatment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiangdong Cheng (Other)
Responsible Party: Sponsor-Investigator, Xiangdong Cheng, Secretary of the party committee, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-GasC-QIBA-1001
Record Dates: First submitted 2024-12-28; First posted 2025-01-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancers; Esophagogastric Junction Cancers
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 combined with SOX (Experimental): QL1706 + SOX (3 cycles) before surgery → radical surgery (D2) → QL1706 + SOX (5 cycles) after surgery → QL1706 monotherapy maintenance (up to 1 year before and after surgery); Surgery is performed 3 - 6 weeks after the last dose of neoadjuvant therapy, and postoperative adjuvant therapy is initiated at least 4 weeks and up to 6 weeks after surgery.
  Phase 1 (initial dose cohort) ： QL1706 5mg/kg ；Phase 1 (dose escalation cohort)：QL1706 7.5mg/kg ；Phase 2：QL1706 RP2D
  Interventions: Drug: QL1706 combined with SOX

INTERVENTIONS:
Drug: QL1706 combined with SOX — QL1706 + SOX (3 cycles) before surgery → radical surgery (D2) → QL1706 + SOX (5 cycles) after surgery → QL1706 monotherapy maintenance （up to 1 year before and after surgery); Phase 1 (initial dose cohort) ： QL1706 5mg/kg ；Phase 1 (dose escalation cohort)：QL1706 7.5mg/kg ；Phase 2：QL1706 RP2D

SUMMARY:
This is a single-center, single-arm clinical study to evaluate the efficacy and safety of QL1706 combined with SOX for the treatment of resectable locally advanced gastric or gastroesophageal junction adenocarcinoma.

The study consists of the following two phases:

Phase 1: The safety introduction phase of QL1706 combined with SOX, using a 3+3 design, enrolled about 6 to 12 patients with locally advanced gastric/gastroesophageal junction adenocarcinoma (primary clinical stage ≥T3 or N+, M0) and underwent 3-week DLT evaluation.

Phase 2: This phase plans to enroll 42 to 45 patients, using investigator-evaluated pCR as the primary endpoint. QL1706 is administered by intravenous infusion of RP2D as defined in Part 1 starting from cycle 1.

Preoperative QL1706 RP2D combined with SOX (3 cycles) → radical surgery (D2) → postoperative QL1706 RP2D combined with SOX (5 cycles) → postoperative maintenance of QL1706 RP2D (up to 1 year before and after surgery); neoadjuvant therapy Surgery should be performed within 3 to 6 weeks after the last dosing, with a minimum interval of 4 weeks after surgery and a maximum interval of 6 weeks recommended for postoperative adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent to join the study voluntarily;
2. Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction;
3. Adenocarcinoma of the stomach or gastroesophageal junction was evaluated by CT/MRI (primary clinical stage ≥T3 or N+, M0, according to AJCC 8th edition staging), including Siewert type II and III tumors
4. Age 18-75 years old, male or female;
5. ECOG PS 0-1 ;
6. Have not received any anti-tumor treatment for gastric or gastroesophageal junction adenocarcinoma, including radiotherapy, chemotherapy, surgery, etc.;
7. Surgical treatment is planned after the completion of neoadjuvant therapy, and R0 resection is expected;
8. Expected survival ≥6 months;
9. Normal functioning of major organs, including:

   1. Blood routine examination (no blood component, cell growth factor are allowed within 7 days before the first use of the study drug) :

      neutrophil count ≥ 1.5×109/L Platelet count ≥ 80×109/L Hemoglobin ≥ 80 g/L
   2. Blood biochemical examination:

      Total bilirubin ≤ 1.5 x ULN ALT ≤ 2.5 x ULN, AST ≤ 2.5 x ULN, Serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 50 mL/min (Cocheroft-Gault formula)
   3. Coagulation function:

   International Standardized ratio (INR) ≤ 1.5 x ULN Activated partial thromboplastin time (APTT) ≤ 1.5 x ULN
10. Fertile female subjects are required to take a serum or urine pregnancy test that is negative within 72 hours prior to the start of the study drug administration, and to use effective contraception (such as Iuds, contraceptives, or condoms) during the trial period and for at least 120 days after the last dose; For male subjects whose partner is a fertile woman, they should be surgically sterilized or agree to use effective contraception during the trial and for 120 days after the last dose;
11. The subject have good compliance and cooperated well with the follow-up
12. Agreed to provide tumor tissue samples

Exclusion Criteria:

1. There are unresectable factors, including unresectable tumor causes or unresectable or refused surgery contraindications;
2. Have received or are receiving any of the following treatment:

   1. any radiation therapy, chemotherapy, or immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.) and other anti-tumor drugs;
   2. being treated with immunosuppressive drugs or systemic hormones for immunosuppressive purposes within 2 weeks prior to the initial use of the investigational drug (dose >10mg/ day prednisone or equivalent); In the absence of active autoimmune disease, inhaled or topical steroid use and adrenocortical hormone replacement with doses >10mg/ day of prednisone or equivalent are permitted;
   3. Received live attenuated vaccine within 4 weeks prior to the first use of the investigational drug; If enrolled, subjects must not receive live vaccine during the study period or within 120 days after the last administration of QL1706;
3. Serious infections (CTCAE > Grade 2) occurred within 4 weeks prior to the first use of the study drug, such as severe pneumonia, bacteremia, and infection complications requiring hospitalization; Baseline chest imaging indicated active pulmonary inflammation, signs and symptoms of infection within 14 days prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, except in cases of prophylactic antibiotic use;
4. Patients with active autoimmune disease requiring systemic treatment within 2 years prior to initial use of the investigational drug or a history of autoimmune disease with recurrence possible [including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (which can be controlled by hormone replacement therapy alone) Patients can be enrolled)];
5. A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation;
6. There are clinical symptoms or diseases of heart that are not well controlled, including but not limited to: (1) NYHA grade II or above heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) Clinically significant supraventricular or ventricular arrhythmias that are not well controlled without or after clinical intervention; (5) QTc> 450ms (male); QTc > 470ms (female);
7. Patients found to have active pulmonary tuberculosis infection through medical history or CT examination, or had a history of active pulmonary tuberculosis infection within 1 year before enrollment, or had a history of active pulmonary tuberculosis infection more than 1 year ago without formal treatment;
8. There are factors that increase the risk of prolonged QTc and abnormal heart rate, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, sudden unexplained death of immediate family members under 40 years of age, or prolonged QT interval accompanied by medication;
9. Active hepatitis (Hepatitis B reference: HBsAg positive and HBV DNA≥2000 IU/ml; Hepatitis C reference: HCV antibody positive and HCV copy number > upper limit of normal);
10. Defined as ≥ grade 2 peripheral neuropathy according to NCI-CTCAE v5.0 standards;
11. Have been diagnosed with other malignancies within 5 years prior to initial dosing, unless malignancies with a low risk of metastasis or death (5-year survival > 90%), such as well-treated basal cell or squamous cell skin cancer of the skin or cervical carcinoma in situ may be considered for inclusion;
12. Known history of severe hypersensitivity to other monoclonal antibodies; Patients with a known history of allergy or hypersensitivity to QL1706, oxaliplatin, and Tigor or any of their components;
13. Known deficiency of dihydropyrimidine dehydrogenase;
14. Upper gastrointestinal obstruction or abnormal physiological function or malabsorption syndrome that may affect the absorption of Tegor;
15. Pregnant or lactating women;
16. Enrolling in another clinical study at the same time, unless it is an observational, non-interventional clinical study or the follow-up period of an interventional study;
17. The investigator determined that there were other factors that might have led to the forced termination of the study, such as other serious medical conditions (including mental illness) requiring co-treatment, alcohol, substance abuse, family or social factors, and factors that might have affected the safety or adhere

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 21 days
Recommended Phase II Dose | 21 days
Pathological complete response | After operation about 2 weeks

SECONDARY OUTCOMES:
major pathological response | After operation about 2 weeks
R0 resection rate | about 15 weeks
ypTNM stage | After operation about 2 weeks
Event-Free Survival | up to approximately 4 years
Disease-Free Survival | approximately 4 years
Overall survival | up to approximately 6 years
Surgery Delay | about 2 months，compared with surgery performed within 3 to 6 weeks after the last administration of neoadjuvant therapy
Incidence and severity of adverse events (including serious adverse events and immune-related adverse events) assessed by CTCAE v5.0 | about 18 months

OTHER OUTCOMES:
Correlation between biomarkers（Such as PD-L1 expression, MMR, EBV and HER2 status） and efficacy（Such as EFS、DFS）） | up to approximately 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
QL1706 + SOX (3 cycles) before surgery → radical surgery (D2) → QL1706 + SOX (5 cycles) after surgery → QL1706 monotherapy maintenance (up to 1 year before and after surgery); Surgery is performed 3 - 6 weeks after the last dose of neoadjuvant therapy, and postoperative adjuvant therapy is initiated at least 4 weeks and up to 6 weeks after surgery.
  Phase 1 (initial dose cohort) ： QL1706 5mg/kg ；Phase 1 (dose escalation cohort)：QL1706 7.5mg/kg ；Phase 1：QL1706 RP2D
Supporting Information: Study Protocol